CLINICAL TRIAL: NCT04481685
Title: A Double-blind, Randomized, Controlled Trial of ATI-450 in Patients With Moderate-severe COVID-19
Brief Title: A Trial of Aclaris Therapeutics, Inc. (ATI)-450 in Patients With Moderate-severe Novel Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT-2020-ATI-450-COVID-19
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATI-450 (Active Comparator): Treated with 50 mg dose of ATI-450, orally, twice daily for 14 days
  Interventions: Drug: ATI-450
- Placebo (Placebo Comparator): Treated with matched placebo, orally, twice daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATI-450 — 50 mg (as determined from Phase I study) per dose. (100 mg per day). Up to a maximum of 14 days while inpatient. Patients discharged home or transferred to the intensive care unit (ICU) will be discontinued off drug permanently.
  Arms: ATI-450
Drug: Placebo — Placebo pill will be taken twice daily preferably spaced 12 hours apart.
  Arms: Placebo

SUMMARY:
COVID-19 morbidity and mortality has been associated with Cytokine Release Syndrome (CRS) and Acute Respiratory Distress Syndrome (ARDS).

ATI-450 is an oral small molecule MAPKAPK2 (MK2) inhibitor that potently inhibits multiple inflammatory cytokines.

The investigator hypothesizes that MK2 pathway blockade during active COVID-19 infection in hospitalized participants will result in improvement in respiratory-failure free survival.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and be willing to sign the Institutional Review Board (IRB)-approved subject informed consent form (ICF) prior to administration of any study-related procedures, or consent from surrogate decision maker when the above criteria cannot be met
* Male or non-pregnant female adult ≥18 years of age at time of enrollment; female patients must have a negative serum pregnancy test at study enrollment
* Has laboratory-confirmed COVID-19 coronavirus infection as determined by polymerase chain reaction (PCR), or other commercial or public health assay in oropharyngeal or nasopharyngeal testing within 14 days of hospitalization. An additional 24-hour COVID-19 PCR test will be performed at KUMC. Patients outside of KUMC will have their samples sent to KUMC as a Central Lab for test processing
* Hospitalized as a result of symptoms and signs related to COVID-19 infection, and ≤14 days since positive test
* Evidence of hypoxic respiratory failure: SpO2≤93% on room air, or SpO2 >93% requiring ≥ 2 Liters (L) O2, or Pa02/Fi02 ratio <300 Millimeter of Mercury (mmHg), or tachypnea (respiratory rate > 30 breaths/min)
* Evidence of pulmonary involvement by: chest imaging or pulmonary exam
* Previous use of hydroxychloroquine or chloroquine is allowed in this study
* Adequate organ function per laboratory tests
* Females of child-bearing potential and males with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for 30 Days for females and 90 days for males following completion of therapy

Exclusion Criteria:

* Known hypersensitivity to ATI-450
* History or evidence of active or latent tuberculosis or recent exposure (within last 30d) to a person with active Tb
* Evidence of active, untreated bacterial infection. Patients who are treated with antibiotics for at least 72 hours, will become eligible for rescreening for trial enrollment
* Active use of immunosuppressant medication(s) (i.e. anti-rejection ,immunomodulators or immunosuppressant drugs, including but not limited to IL-6 inhibitors, TNF inhibitors, anti-IL-1 agents and Janus kinase (JAK) inhibitors within 5 half-lives or 30 days (whichever is longer) prior to randomization. (Use of hydroxychloroquine/chloroquine should be discontinued)
* Oncology patients who are on active chemotherapy or immunotherapy. However, oncology patients who come off active therapy prior to enrollment and have absolute neutrophil count (ANC) ≥1500/mmc are eligible for enrollment
* Active participation in a concurrent COVID-19 clinical trial with investigative medical drug therapies. However, co-enrollment for non-investigative drug therapies will be allowed; use or re-purposing of FDA approved treatments will be considered at the discretion of the medical monitor
* In the opinion of the investigator, unlikely to survive for at least 48 hours from screening or anticipate mechanical ventilation within 48 hours
* Pregnancy or breast feeding
* Prisoner
* Intubation and ventilation at time of enrollment
* Known history for HIV, hepatitis B or C infection. Patients with serologic evidence of hepatitis B vaccination (hepatitis B surface antibody without the presence of hepatitis B surface antigen) will be allowed to participate
* History of a past or current medical condition that in the opinion of the treating physician would compromise patient safety (e.g. uncontrolled HIV) by participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Gan, MD, PhD, Principal Investigator — The University of Kansas; Deepika Polineni, MD, PhD, Principal Investigator — The University of Kansas
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATI-450 | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATI-450 | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 10 | 16
  >=65 years | 4 | 0 | 4
Age, Continuous [Median (Full Range); unit: years] | 64 [34 to 85] | 63 [43 to 67] | 63 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 6 | 12
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Failure-free Survival in Participants With Moderate-severe COVID-19 Who Are Treated With ATI-450
Description: Proportion of responders on Day 14 defined as all subjects who are alive, free of respiratory failure (do not require supplemental oxygen) and do not experience negative intercurrent events by Day 14 of the trial will be considered responders, as assessed by participant medical records.
Time Frame: Study day 14
Measure: Number (90% Confidence Interval); unit: percentage of total patients
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
percentage of total patients | 50 [22.2 to 77.8] | 60 [30.4 to 85]

2. Secondary Outcome: Change in 7 Point-ordinal Scale
Description: Using World Health Organization (WHO) COVID-19 Ordinal scale measuring: Participants were assessed on a 7-point categorical scale, and change in scores between timepoints is reported. This scale measures illness severity over time and has a range of 0-7.
  * 0- Uninfected: No clinical or virological evidence of infection.
  * 1- Ambulatory: No limitation of activities.
  * 2- Ambulatory: Limitation of activities.
  * 3- Hospitalized, mild disease: Hospitalized, no oxygen.
  * 4- Hospitalized, mild disease: Oxygen by mask or nasal prongs.
  * 5- Hospitalized, severe disease: Non- invasive ventilation or high- flow oxygen.
  * 6- Hospitalized, severe disease: Intubation and mechanical ventilation.
  * 7- Hospitalized, severe disease: Ventilation + organ support; pressors, Renal Replacement Therapy (RRT), Extracorporeal Membrane Oxygenation (ECMO).
Time Frame: Baseline, Day 7, Day 14, Day 28 and follow-up up to 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline to Day 7 | 0 (0.4714) | 0 (0.4714)
  baseline to EoT | 0.7 (1.2517) | 0.1 (1.3703)
  baseline to Day 14 | 1.7 (1.5670) | 1.9 (1.7920)
  baseline to Day 28 | 2.7 (1.1738) | 2.2 (0.9189)

3. Secondary Outcome: Number of Participants With a Need for Advanced Respiratory Care
Description: Derived from medical record
Time Frame: Baseline and continuous throughout hospitalization up to 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 2 | 1

4. Secondary Outcome: All-cause Mortality
Description: Noted in participant medical record
Time Frame: Baseline and through day 60
Measure: Number; unit: participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
participants | 1 | 1

5. Secondary Outcome: Treatment-emergent Adverse Events
Description: Number of adverse events (AEs), as assessed by CTCAE v5.0.
  Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL (Activities of Daily Living).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to Day 60
Measure: Number; unit: adverse events
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
adverse events
  Any Grade | 14 | 6
  Grade 1-2 | 12 | 6
  Grade 3 | 2 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

6. Secondary Outcome: Treatment-emergent Serious Adverse Events
Description: Number of serious adverse events (SAEs), as assessed by CTCAE v5.0.
  Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to Day 60
Population: Report of any treatment-emergent Serious adverse events (TeSAE)
Measure: Number; unit: serious adverse events
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
serious adverse events
  Any Grade | 2 | 2
  Grade 1 or 2 | 0 | 1
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Grade 5 | 1 | 1

7. Secondary Outcome: Number of Participants With Normalization of Fever for 24 Hours
Description: Standard daily temperature measurement and obtained from participant medical record
Time Frame: Baseline through day 14 or at discharge <day 14
Measure: Number; unit: participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
participants | 9 | 9

8. Secondary Outcome: Number of Participants Who Develop New Bacterial Infection
Description: Noted in participant medical record
Time Frame: Continuous throughout hospitalization up to 14 days
Measure: Number; unit: participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
participants | 0 | 0

9. Secondary Outcome: Number of Participants Who Develop New Fungal Infection
Description: Noted in participant medical record
Time Frame: Continuous throughout hospitalization up to 14 days
Measure: Number; unit: participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
participants | 1 | 0

10. Secondary Outcome: Number of Adult Respiratory Distress Syndrome (ARDS2)
Description: Noted in participant medical record
Time Frame: From day 1 though day 14 or at discharge <day 14
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1

11. Secondary Outcome: Change in Serum Cytokine Interleukin (IL)-6
Description: Plasma was assayed by Confluence Discovery Technologies using the MesoScale Discovery Platform from biobanked samples stored from the University of Kansas Medical Center (KUMC) Biobanking and Biomarker Validation (BBV) Core, expressed in pg/mL. Change in biomarker was reported as a percent based on (EOT or D14)/baseline x100%.
Time Frame: Baseline to End of Treatment, or Day 14
Population: baseline vs EoT
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
percentage of baseline | 34.8 [30.6 to 41.3] | 137.6 [16.5 to 187]

12. Secondary Outcome: Change in Serum Cytokine IL-8
Description: as for outcome 11
Time Frame: Baseline to End of Treatment, or Day 14
Population: baseline vs EoT
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
percentage of baseline | 40.1 [23.4 to 74.1] | 82.3 [69.1 to 145.5]

13. Secondary Outcome: Change in Serum Cytokines IL-1β
Description: as for outcome 11
Time Frame: Baseline to End of Treatment, or Day 14
Population: Baseline vs EoT - this could not be measured because analyte could not be detected
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
percentage of baseline | NA (NA) — Baseline vs EoT - this could not be measured because analyte could not be detected | NA (NA) — Baseline vs EoT - this could not be measured because analyte could not be detected

14. Secondary Outcome: Change in Serum Cytokine Tumor Necrosis Factor (TNF-α)
Description: as for outcome 11
Time Frame: Baseline to End of Treatment, or Day 14
Population: baseline vs EoT
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | ATI-450 | Placebo
Number analyzed (Participants) | 10 | 10
percentage of baseline | 56.6 [32.1 to 119.5] | 104.1 [85.4 to 134.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from initiation of study treatment and continues until the Day 60 safety follow-up.
Description: Per protocol, medical history adverse events are recorded and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Serious adverse event and adverse event monitoring begins after initiation of study treatment and continues until the Day 60 safety follow-up. This Day 60 follow-up check and will be done by phone.
Arm/Group | ATI-450 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/10
Other Adverse Events (participants affected / at risk) | 7/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-450 (N=10) | Placebo (N=10)
multi-organ failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-450 (N=10) | Placebo (N=10)
superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
cardiac troponin (Cardiac disorders) | 1 (1) | 0 (0)
lymphocele (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
GGT increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
aspartate aminotransferase increase (Hepatobiliary disorders) | 2 (2) | 0 (0)
alanine aminotransferase increase (Hepatobiliary disorders) | 2 (2) | 0 (0)
creatinine increased (Renal and urinary disorders) | 1 (1) | 0 (0)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
non-cardiac chest pain (Cardiac disorders) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
thrush (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT04481685/Prot_002.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT04481685/SAP_003.pdf